CLINICAL TRIAL: NCT00359424
Title: Interventional Management of Stroke Trial (IMS III): A Phase III Clinical Trial Examining Whether a Combined Intravenous (IV) and Intra-Arterial (IA) Approach to Recanalization is Superior to Standard IV Rt-PA (Activase®) Alone
Brief Title: Interventional Management of Stroke (IMS) III Trial
Acronym: IMSIII
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: NINDS/NIH-DSMB recommended halting trial due to futility, no safety concerns.
Sponsor: Joseph Broderick (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medical University of South Carolina (Other); University of Calgary (Other)
Responsible Party: Sponsor-Investigator, Joseph Broderick, Professor and Chairman Department of Neurology, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01NS052220 (NIH); U01NS052220 (NIH); U01NS054630 (NIH); 2009-017454-12 (EudraCT Number)
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Stroke
Keywords: acute ischemic stroke; rt-PA; thrombolytic; recombinant tissue plasminogen activator; recanalization; blood clot; stroke; clot-dissolving; Activase®; Actilyse®; Concentric Merci® Retriever; EKOS® Micro-Infusion catheter (MicroLysus); The Penumbra System™; Standard microcatheter
MeSH Terms: conditions — Stroke; Ischemic Stroke; Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous (IV) rt-PA alone (Active Comparator): Group one will receive the standard dose of intravenous (IV) rt-PA alone given over an hour.
  Interventions: Drug: IV rt-PA alone
- Endovascular therapy (Experimental): Group two will receive a lower dose or a standard dose of IV rt-PA and then undergo an angiogram test (cerebral angiography) right after the medicine is given to check for blood clots. If a clot is not seen then no more treatment will be given. If a clot is seen, the neurointerventionalist will then choose (based on the location and extent of the blood clot) a protocol approved endovascular treatment given directly in the brain artery that will be most effective in reopening the blocked artery.
  Interventions: Drug: IV rt-PA alone; Other: endovascular therapy

INTERVENTIONS:
Drug: IV rt-PA alone — Intravenous (IV) recombinant tissue plasminogen activator (rt-PA) is the only approved acute stroke therapy; Group one will receive the standard dose of IV rt-PA given over an hour.
  Other Names: Activase®, Actilyse®
Other: endovascular therapy — Group two will receive a lower dose or the standard dose of IV rt-PA and then undergo an angiogram test (cerebral angiography) right after the medicine is given to check for blood clots. If a clot is not seen then no more treatment will be given. If a clot is seen, the neurointerventionalist will then choose a protocol approved endovascular treatment given directly in the brain artery that will be most effective in reopening the blocked artery. Endovascular therapy can be implemented with or without interarterial rt-PA use.
  Other Names: Activase®, Actilyse®
  Arms: Endovascular therapy

SUMMARY:
The purpose of this study is to compare two different treatment approaches to recanalization started within 3 hours of symptom onset-combined intravenous (IV) and endovascular therapy and standard intravenous (IV) rt-PA alone.

DETAILED DESCRIPTION:
Stroke remains a major cause of death and disability. Acute thrombolytic therapy offers the potential to achieve early recanalization (reopening of blocked arteries), save tissues, and improve outcome. Currently, intravenous (IV) recombinant tissue plasminogen activator (rt-PA) is the only approved acute stroke therapy. IV rt-PA is an effective therapy for acute ischemic stroke but has substantial limitations when used alone to open blocked arteries The Interventional Management of Stroke (IMS III) Trial is a multi-center study that will compare two different treatment approaches for restoring blood flow to the brain. One approach, giving the clot-dissolving drug rt-PA, is already FDA-approved when given through a vein (IV). This treatment will be compared to a new approach, giving rt-PA at a lower dose first through IV in the arm and then, if a blood clot in the brain artery is found, through a small tube or catheter at the site of the blood clot (intra-arterial or IA) to see which is better. Both approaches must be initiated within three hours of stroke onset.

The primary goal of this trial is to determine if individuals with ischemic stroke treated with rt-PA using an endovascular therapy approach to recanalization started within 3 hours of onset are more likely to have a better outcome than individuals treated with standard IV rt-PA alone. While information on device use was collected, individual device performance was not a primary outcome.

Nine hundred participants with moderate to severe ischemic stroke will be enrolled at more than 50 centers in the United States, Canada, Australia and Europe.

Subjects will be randomized in a 2:1 ratio to receive endovascular therapy or IV only with adjustment for clinical site and NIHSSS strata. If enrolled under Amendment 5 or later both treatment groups will receive the standard approved therapy dose of rt-PA (0.9 mg/kg, 90 mg max) administered intravenously over one hour. The consent process and randomization can take place prior to or anytime up to forty minutes after the IV bolus dose. If, at the 40 minute time point, no consent has been obtained or randomization has not been completed, the patient will no longer be eligible for IMS III enrollment. After consent, the endovascular therapy group will then undergo immediate angiography. If clot is not demonstrated, no more treatment is administered.

If clot is demonstrated, the neurointerventionalist will then choose from currently available but trial defined endovascular therapy approaches, choosing the treatment they feel will be most effective in attempting to reopen the blocked artery. These approaches utilize local regulatory, US FDA and IMS III Executive Committee approved devices for the intra-arterial infusion of investigational rt-PA using standard microcatheter or the EKOS Micro-Infusion Catheter® (in US) or embolectomy devices including the Concentric Retriever Device®, the Penumbra System ™, or the Solitaire™ FR Revascularization Device. All devices must be used per the manufacturer's instructions for use. Endovascular therapy, whether initially with the Merci® Retriever, EKOS Micro-Infusion Catheter, Penumbra System™, Solitaire™, a future device, or infusion of IA rt-PA via a standard microcatheter, must be started within 5 hours and completed within 7 hours of symptom onset. The maximum dose of IA rt-PA is 22mg (maximum 2 to 4 mg bolus and infusion at a rate of 10 mg/hr). Use of tandem devices (i.e. EKOS Micro-Infusion Catheter, Merci Retriever®, Penumbra System™, or Solitaire™) in a single case is a protocol violation. Only standard microcatheter rt-PA infusion therapy may be administered following attempt with a device.

The primary measure of benefit in this trial is the ability of the individual with stroke to live and function independently 3 months after the stroke. This trial will also determine and compare the safety and cost effectiveness of the combined endovascular therapy to the standard IV rt-PA approach.

Duration of the study for participants is approximately 12 months.

ELIGIBILITY:
Inclusion Criteria

* Age: 18 through 82 years (i.e., candidates must have had their 18th birthday, but not had their 83rd birthday)
* Initiation of intravenous rt-PA within 3 hours of onset of stroke symptoms. Time of onset is defined as the last time when the subject was witnessed to be at baseline (i.e., subjects who have stroke symptoms upon awakening will be considered to have their onset at beginning of sleep)
* An NIHSSS >/= 10 at the time that intravenous rt-PA is begun or an NIHSSS >7 and <10 with an occlusion seen in M1, ICA or basilar artery on CTA at institutions where baseline CTA imaging is standard of care for acute stroke patients.
* Investigator verification that the subject has received/ is receiving the correct IV rt-PA dose for the estimated weight prior to randomization

Exclusion Criteria

* History of stroke in the past 3 months
* Previous intra-cranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arteriovenous malformation
* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT scan is normal
* Hypertension at time of treatment; systolic BP > 185 or diastolic > 110 mm Hg) or aggressive measures to lower BP to below these limits are needed.
* Presumed septic embolus, or suspicion of bacterial endocarditis
* Presumed pericarditis, including pericarditis after acute MI
* Suspicion of aortic dissection
* Recent (within 30 days) surgery or biopsy of parenchymal organ
* Recent (within 30 days) trauma, with internal injuries or ulcerative wounds
* Recent (within 90 days) severe head trauma or head trauma with loss of consciousness
* Any active or recent (within 30 days) hemorrhage
* Pts with known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency or oral anticoagulant therapy require coagulation labs results prior to enrollment. Any subject with INR > 1.7 or institutionally equivalent prothrombin time is excluded. Patients without history or suspicion of coagulopathy do not require INR or prothrombin time lab results to be available prior to enrollment.
* Females of childbearing potential who are known to be pregnant and/or lactating or who have positive pregnancy tests on admission
* Baseline lab values: glucose < 50 mg/dl or > 400 mg/dl, platelets <100,000, or Hct <25
* Requires hemodialysis or peritoneal dialysis, or has a contraindication to an angiogram for whatever reason
* Received heparin or a direct thrombin inhibitor (Angiomax, argatroban, Refludan, Pradaxa) within 48 hours must have a normal partial thromboplastin time (PTT) to be eligible
* History of an arterial puncture at a non-compressible site or a lumbar puncture in the previous 7 days
* History of seizure at onset of stroke
* History of a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, mRS score at baseline must be < 2. This excludes patients who live in a nursing home or who are not fully independent for activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.)
* Other serious, advanced, or terminal illness
* Any other condition that the investigator feels would pose a significant hazard to the subject if Activase (Alteplase) therapy is initiated
* Current participation in another research drug treatment protocol
* Informed consent is not or cannot be obtained.
* High density lesion consistent with hemorrhage of any degree on baseline imaging
* Significant mass effect with midline shift on baseline imaging
* Large (>1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan. (ASPECTS of < 4 can be used as a guideline) Sulcal effacement and/or loss of grey-white differentiation are not contraindications to tx
* CT evidence of intrapararenchymal tumor
* Baseline CTA without evidence of arterial occlusion

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2006-08; Primary Completion 2012-07 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P. Broderick, MD, Principal Investigator — Primary Neurologist Investigator, University of Cincinnati Academic Health Center; Thomas A. Tomsick, MD, Principal Investigator — Primary Interventional Investigator, University of Cincinnati Academic Health Center
Locations (71):
- United States (49):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Barrow Neurology Clinics at St. Joseph's Hospital and Medical Center, 222 W. Thomas Road, Suite 404, Phoenix, Arizona
  - Mayo Clinic Arizona, 5777 E. Mayo Blvd., Scottsdale, Arizona
  - UCLA Medical Center, 924 Westwood Blvd., Suite 300, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Santa Monica-UCLA Medical Center, 1250 16th Street, Santa Monica, California
  - Colorado Neurological Institute, Swedish Medical Center, 501 E. Hampden Ave., Englewood, Colorado
  - Stroke Center at Hartford, 80 Seymour St. Rm JB603, Hartford, Connecticut
  - Morton Plant Mease Health Care, 300 Pinellas Street MS 49, Clearwater, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Alexian Brothers Medical Center, 800 Biesterfield Rd., Elk Grove Village, Illinois
  - Ruan Neurological Mercy Medical Center, 1111 6th Ave., Ste. 400, Des Moines, Iowa
  - St. Elizabeth Medical Center South, One Medical Village Drive, Edgewood, Kentucky
  - St Luke's West Hospital, 7380 Turfway Rd., Florence, Kentucky
  - St. Luke's Hospital East, 85 N. Grand Ave., Fort Thomas, Kentucky
  - University of Louisville, Kentucky Neuroscience Research, Stroke Research, 401 East Chestnut Street, Suite 520, Louisville, Kentucky
  - Johns Hopkins University, 1500 Orleans St. 3M South, Baltimore, Maryland
  - Massachusetts General Hospital, 55 Fruit Street, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, 2799 W Grand Blvd, CFP-260, Detroit, Michigan
  - Michigan State University, Sparrow Hospital, B 401 Clinical Center, East Lansing, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University/Barnes Jewish Hospital, 660 S. Euclid Avenue, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Suny Upstate Medical University, Syracuse, New York
  - Mission Hospital, 509 Biltmore Avenue, Asheville, North Carolina
  - University of North Carolina, CB # 7025, 7003 Neurosciences Hospital, 7th Floor, Chapel Hill, North Carolina
  - The Christ Hospital, 2139 Auburn Ave., Cincinnati, Ohio
  - The University Hospital, 234 Goodman Ave., Cincinnati, Ohio
  - Good Samaritan Hospital, 375 Dixmyth Ave., Cincinnati, Ohio
  - The Jewish Hospital of Cincinnati, 4777 East Galbraith Rd, Cincinnati, Ohio
  - Mercy Hospital, Western Hills, 3131 Queen City Ave., Cincinnati, Ohio
  - Mercy Hospital, Mt Airy, 2446 Kipling Ave., Cincinnati, Ohio
  - Mercy Hospital Anderson, 7500 State Rd, Cincinnati, Ohio
  - University Hospitals of Cleveland, Case Western Reserve University,Case Western Neurological Unit, 11100 Euclid Avenue, Lakeside 5508, Cleveland, Ohio
  - Riverside Methodist Hospital, 3535 Olentangy River Road, Columbus, Ohio
  - Mercy Hospital Fairfield, 3000 Mack Rd., Fairfield, Ohio
  - Bethesda North Hospital, 10500 Montgomery Rd., Montgomery, Ohio
  - OHSU, Oregon Stroke Center, Providence St. Vincent's Hospital, Providence Portland Hospital, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital Center, 1200 South Cedar Crest Blvd., Allentown, Pennsylvania
  - PENN State M.S. Hershey Medical Center, 500 University Drive MC: HS 86, Long Lane Rom HG:212, Hershey, Pennsylvania
  - Allegheny General Hospital, 420 East North Avenue, East Wing Office Bldg., Suite 206, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Medical Center, 200 Lothrop Street, PUH C-400, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University Medical Center at Brackenridge Hospital, Austin, Texas
  - University of Texas Medical School at Houston, 6431 Fannin, MSB 7.044, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Froedtert Hospital, Medical College of Wisconsin, 9200 W. Wisconsin Avenue, Milwaukee, Wisconsin
- Australia (4):
  - Royal Prince Alfred Hospital, Level 10 King George V Building, Missenden Rd, Camperdown
  - St. Vincent's Hospital, Clincial Trial Centre Level 5, 378 Victoria St., Darlinghurst, Sydney
  - Royal Melbourne Hospital, Dept. of Neurology, 4 East, Grattan St, Parkville, Victoria
  - Monash Medical Center, Dept. of Neurology, 246 Clayton Rd, Clayton, Victoria
- Canada (7):
  - University of Calgary, Calgary Health Region/Foothills Hospital, 1403 29th Street NW, Calgary, Alberta
  - University of British Columbia, Vancouver General Hospital, VGH Stroke Program, Gordon & Leslie Diamond Healthcare Centre, 2775 Laurel St., 8th Fl., Ste. 8295, Vancouver, British Columbia
  - The Ottawa Hospital, Civic Campus, CPC Main, RM 36, Box 608, 1053 Carling Avenue, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, 5th Floor Rm. 447, 399 Bathurst St., Toronto, Ontario
  - Centre Hospital University of Montreal, Montreal, Quebec
- Bichat Stroke Centre, Paris, Cedex, France
- Germany (5):
  - Technische Universität, Dresden, Dresden
  - University of Freiburg, Freiburg im Breisgau
  - Ernst Moritz Arndt University, Greifswald
  - Martin-Luther University, Halle
  - Asklepios Klinik Nord Heidberg, Hamburg
- St. Antonius Hospital, Nieuwegein, Netherlands
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Vall d´Hebron, Barcelona
- Switzerland (2):
  - University Hospital Basel, Basel
  - Centre Hospitalier, University Vaudois, Lausanne

REFERENCES:
- [Derived] van der Ende NAM, den Hartog SJ, Broderick JP, Khatri P, Visser-Meily JMA, van Leeuwen N, Lingsma HF, Roozenbeek B, Dippel DWJ; IMS III Investigators. Disentangling the Association Between Neurologic Deficits, Patient-Reported Impairments, and Quality of Life After Ischemic Stroke. Neurology. 2023 Mar 28;100(13):e1321-e1328. doi: 10.1212/WNL.0000000000206747. Epub 2023 Jan 4. PMID 36599699
- [Derived] van der Ende NA, Roozenbeek B, Broderick JP, Khatri P, Lingsma HF, Dippel DW. Blinding of outcome assessors and its association with outcome in a randomized open-label stroke trial. Int J Stroke. 2023 Jun;18(5):562-568. doi: 10.1177/17474930221131706. Epub 2022 Oct 19. PMID 36169032
- [Derived] Chalos V, van der Ende NAM, Lingsma HF, Mulder MJHL, Venema E, Dijkland SA, Berkhemer OA, Yoo AJ, Broderick JP, Palesch YY, Yeatts SD, Roos YBWEM, van Oostenbrugge RJ, van Zwam WH, Majoie CBLM, van der Lugt A, Roozenbeek B, Dippel DWJ; MR CLEAN Investigators. National Institutes of Health Stroke Scale: An Alternative Primary Outcome Measure for Trials of Acute Treatment for Ischemic Stroke. Stroke. 2020 Jan;51(1):282-290. doi: 10.1161/STROKEAHA.119.026791. Epub 2019 Dec 4. PMID 31795895
- [Derived] Simpson KN, Simpson AN, Mauldin PD, Palesch YY, Yeatts SD, Kleindorfer D, Tomsick TA, Foster LD, Demchuk AM, Khatri P, Hill MD, Jauch EC, Jovin TG, Yan B, von Kummer R, Molina CA, Goyal M, Schonewille WJ, Mazighi M, Engelter ST, Anderson C, Spilker J, Carrozzella J, Ryckborst KJ, Janis LS, Broderick JP; Interventional Management of Stroke (IMS) III Investigators. Observed Cost and Variations in Short Term Cost-Effectiveness of Therapy for Ischemic Stroke in Interventional Management of Stroke (IMS) III. J Am Heart Assoc. 2017 May 8;6(5):e004513. doi: 10.1161/JAHA.116.004513. PMID 28483774
- [Derived] Venema E, Mulder MJHL, Roozenbeek B, Broderick JP, Yeatts SD, Khatri P, Berkhemer OA, Emmer BJ, Roos YBWEM, Majoie CBLM, van Oostenbrugge RJ, van Zwam WH, van der Lugt A, Steyerberg EW, Dippel DWJ, Lingsma HF. Selection of patients for intra-arterial treatment for acute ischaemic stroke: development and validation of a clinical decision tool in two randomised trials. BMJ. 2017 May 3;357:j1710. doi: 10.1136/bmj.j1710. PMID 28468840
- [Derived] Mulder MJ, Venema E, Roozenbeek B, Broderick JP, Yeatts SD, Khatri P, Berkhemer OA, Roos YB, Majoie CB, van Oostenbrugge RJ, van Zwam WH, van der Lugt A, Steyerberg EW, Dippel DW, Lingsma HF. Towards personalised intra-arterial treatment of patients with acute ischaemic stroke: a study protocol for development and validation of a clinical decision aid. BMJ Open. 2017 Mar 22;7(3):e013699. doi: 10.1136/bmjopen-2016-013699. PMID 28336740
- [Derived] Broderick JP, Berkhemer OA, Palesch YY, Dippel DW, Foster LD, Roos YB, van der Lugt A, Tomsick TA, Majoie CB, van Zwam WH, Demchuk AM, van Oostenbrugge RJ, Khatri P, Lingsma HF, Hill MD, Roozenbeek B, Jauch EC, Jovin TG, Yan B, von Kummer R, Molina CA, Goyal M, Schonewille WJ, Mazighi M, Engelter ST, Anderson CS, Spilker J, Carrozzella J, Ryckborst KJ, Janis LS, Simpson KN; IMS III Investigators; MR CLEAN Investigators. Endovascular Therapy Is Effective and Safe for Patients With Severe Ischemic Stroke: Pooled Analysis of Interventional Management of Stroke III and Multicenter Randomized Clinical Trial of Endovascular Therapy for Acute Ischemic Stroke in the Netherlands Data. Stroke. 2015 Dec;46(12):3416-22. doi: 10.1161/STROKEAHA.115.011397. Epub 2015 Oct 20. PMID 26486865
- [Derived] Abou-Chebl A, Yeatts SD, Yan B, Cockroft K, Goyal M, Jovin T, Khatri P, Meyers P, Spilker J, Sugg R, Wartenberg KE, Tomsick T, Broderick J, Hill MD. Impact of General Anesthesia on Safety and Outcomes in the Endovascular Arm of Interventional Management of Stroke (IMS) III Trial. Stroke. 2015 Aug;46(8):2142-8. doi: 10.1161/STROKEAHA.115.008761. Epub 2015 Jul 2. PMID 26138125
- [Derived] Al-Ali F, Elias JJ, Tomsick TA, Liebeskind DS, Broderick JP; IMS Study Groups. Relative Influence of Capillary Index Score, Revascularization, and Time on Stroke Outcomes From the Interventional Management of Stroke III Trial. Stroke. 2015 Jun;46(6):1590-4. doi: 10.1161/STROKEAHA.115.009066. Epub 2015 May 7. PMID 25953374
- [Derived] Palesch YY, Yeatts SD, Tomsick TA, Foster LD, Demchuk AM, Khatri P, Hill MD, Jauch EC, Jovin TG, Yan B, von Kummer R, Molina CA, Goyal M, Schonewille WJ, Mazighi M, Engelter ST, Anderson C, Spilker J, Carrozzella J, Ryckborst KJ, Janis LS, Simpson A, Simpson KN, Broderick JP; Interventional Management of Stroke III Investigators. Twelve-Month Clinical and Quality-of-Life Outcomes in the Interventional Management of Stroke III Trial. Stroke. 2015 May;46(5):1321-7. doi: 10.1161/STROKEAHA.115.009180. Epub 2015 Apr 9. PMID 25858239
- [Derived] Menon BK, Qazi E, Nambiar V, Foster LD, Yeatts SD, Liebeskind D, Jovin TG, Goyal M, Hill MD, Tomsick TA, Broderick JP, Demchuk AM; Interventional Management of Stroke III Investigators. Differential Effect of Baseline Computed Tomographic Angiography Collaterals on Clinical Outcome in Patients Enrolled in the Interventional Management of Stroke III Trial. Stroke. 2015 May;46(5):1239-44. doi: 10.1161/STROKEAHA.115.009009. Epub 2015 Mar 19. PMID 25791716
- [Derived] Tomsick TA, Yeatts SD, Liebeskind DS, Carrozzella J, Foster L, Goyal M, von Kummer R, Hill MD, Demchuk AM, Jovin T, Yan B, Zaidat OO, Schonewille W, Engelter S, Martin R, Khatri P, Spilker J, Palesch YY, Broderick JP; IMS III Investigators. Endovascular revascularization results in IMS III: intracranial ICA and M1 occlusions. J Neurointerv Surg. 2015 Nov;7(11):795-802. doi: 10.1136/neurintsurg-2014-011318. Epub 2014 Oct 23. PMID 25342652
- [Derived] Simpson KN, Simpson AN, Mauldin PD, Hill MD, Yeatts SD, Spilker JA, Foster LD, Khatri P, Martin R, Jauch EC, Kleindorfer D, Palesch YY, Broderick JP; IMS III Investigators. Drivers of costs associated with reperfusion therapy in acute stroke: the Interventional Management of Stroke III Trial. Stroke. 2014 Jun;45(6):1791-8. doi: 10.1161/STROKEAHA.113.003874. Epub 2014 May 13. PMID 24876261
- [Derived] Goyal M, Almekhlafi MA, Fan L, Menon BK, Demchuk AM, Yeatts SD, Hill MD, Tomsick T, Khatri P, Zaidat OO, Jauch EC, Eesa M, Jovin TG, Broderick JP. Evaluation of interval times from onset to reperfusion in patients undergoing endovascular therapy in the Interventional Management of Stroke III trial. Circulation. 2014 Jul 15;130(3):265-72. doi: 10.1161/CIRCULATIONAHA.113.007826. Epub 2014 May 9. PMID 24815501
- [Derived] Yeatts SD, Martin RH, Coffey CS, Lyden PD, Foster LD, Woolson RF, Broderick JP, Di Tullio MR, Jungreis CA, Palesch YY; IMS III Investigators. Challenges of decision making regarding futility in a randomized trial: the Interventional Management of Stroke III experience. Stroke. 2014 May;45(5):1408-14. doi: 10.1161/STROKEAHA.113.003925. Epub 2014 Apr 3. PMID 24699059
- [Derived] Liebeskind DS, Tomsick TA, Foster LD, Yeatts SD, Carrozzella J, Demchuk AM, Jovin TG, Khatri P, von Kummer R, Sugg RM, Zaidat OO, Hussain SI, Goyal M, Menon BK, Al Ali F, Yan B, Palesch YY, Broderick JP; IMS III Investigators. Collaterals at angiography and outcomes in the Interventional Management of Stroke (IMS) III trial. Stroke. 2014 Mar;45(3):759-64. doi: 10.1161/STROKEAHA.113.004072. Epub 2014 Jan 28. PMID 24473178
- [Derived] Hill MD, Demchuk AM, Goyal M, Jovin TG, Foster LD, Tomsick TA, von Kummer R, Yeatts SD, Palesch YY, Broderick JP; IMS3 Investigators. Alberta Stroke Program early computed tomography score to select patients for endovascular treatment: Interventional Management of Stroke (IMS)-III Trial. Stroke. 2014 Feb;45(2):444-9. doi: 10.1161/STROKEAHA.113.003580. Epub 2013 Dec 12. PMID 24335227
- [Derived] Broderick JP, Palesch YY, Demchuk AM, Yeatts SD, Khatri P, Hill MD, Jauch EC, Jovin TG, Yan B, Silver FL, von Kummer R, Molina CA, Demaerschalk BM, Budzik R, Clark WM, Zaidat OO, Malisch TW, Goyal M, Schonewille WJ, Mazighi M, Engelter ST, Anderson C, Spilker J, Carrozzella J, Ryckborst KJ, Janis LS, Martin RH, Foster LD, Tomsick TA; Interventional Management of Stroke (IMS) III Investigators. Endovascular therapy after intravenous t-PA versus t-PA alone for stroke. N Engl J Med. 2013 Mar 7;368(10):893-903. doi: 10.1056/NEJMoa1214300. Epub 2013 Feb 7. PMID 23390923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 656 participants underwent randomization
  * participants to endovascular therapy >> and 222 to intravenous t-PA alone) at 58 study >> centers between August 25, 2006, and April 17, >> 2012 in the United States (41 sites), Canada (7), >> Australia (4), and Europe (6)
Groups:
- Endovascular Therapy: Endovascular therapy (group two) received a lower dose (0.09mg per kg bolus and 0.54mg/kilogram infusion over 40 minutes, maximum dose 53.6mg) or after Amendment #5, a standard dose of IV rt-PA (.9mg/kg with 10% as a bolus and the remainder over one hour) and then underwent an angiogram test (cerebral angiography) right after the medicine was given to check for blood clots. If a clot was not seen, then no more treatment was given. If a clot was seen, the neurointerventionalist chose (based on the location and extent of the blood clot) a protocol approved endovascular treatment given directly in the brain artery that would be most effective in reopening the blocked artery.
- IV Rt-PA Alone: IV rt-PA alone (group one) received the standard dose (.9mg per kilogram with 10% as a bolus and the remainder as an infusion over 1 hour -maximum dose 90mg) of intravenous (IV) rt-PA alone.
Period: Overall Study
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Started | 434 | 222
90 Day Follow up | 343 | 172
180 Day Follow up | 325 | 167
270 Day Follow up | 313 | 159
Completed | 304 | 155
Not Completed | 130 | 67
Not completed — Death | 99 | 58
Not completed — Lost to Follow-up | 19 | 7
Not completed — Withdrawal by Subject | 10 | 2
Not completed — follow up not conducted | 2 | 0

BASELINE CHARACTERISTICS:
Population: A sample of 900 was calculated to provide an effect size of 10 percentage points assuming that 40% of the patients had a good outcome in the IV t-PA group, as noted in patients in the NINDS rt-PA Stroke Study who had age and baseline stroke severity similar to the eligibility criteria for the IMS3 trial. The trial was halted at 656 subjects.
Groups:
- IV Rt-PA Alone: Group one will receive the standard dose of intravenous (IV) rt-PA alone given over an hour.
- Total: Total of all reporting groups
Arm/Group | Endovascular Therapy | IV Rt-PA Alone | Total
Number analyzed (Participants) | 434 | 222 | 656
Age, Continuous [Median (Full Range); unit: years] | 69 [23 to 89] | 68 [23 to 84] | 69 [23 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 100 | 316
  Male | 218 | 122 | 340
NIHSS Score [Median (Full Range); unit: Score on a scale] — The National Institutes of Health Stroke Scale (NIHSS), a serial measure of neurologic deficit, is a 42-point scale that >> quantifies neurologic deficits in 11 categories, with 0 indicating normal function without neurologic deficit and higher
  >> scores indicating greater severity of deficit.
  Score on a scale | 17 [7 to 40] | 16 [8 to 30] | 17 [7 to 40]
Time from stroke onset to initiation of IV rt-PA [Mean (Standard Deviation); unit: minutes] — Time from stroke onset to initiation of intravenous (IV) rt-PA in minutes.
  minutes | 122.4 (33.7) | 121.2 (33.8) | 122.0 (33.7)
NIHSS Score Strata [Number; unit: participants]
  NIHSS Score <20 | 302 | 150 | 452
  NIHSS Score > = 20 | 132 | 72 | 204

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Scale (mRS) Score Dichotomized to 0-2 Versus Greater Than 2.
Description: The modified Rankin Scale (mRS) runs from 0-6 running from perfect health without symptoms to death. 0 - No symptoms at all. 1 - No significant disability. Able to carry out all usual duties and activities. 2 - Slight disability. Unable to carry out all previous activities but able to look after own affairs without assistance. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to walk unassisted and unable to attend to own bodily needs without assistance. 5 - Severe disability. Bedridden, incontinent, and requires constant nursing care and attention. 6 - Dead. Persons with a Rankin of 0-2 are considered functionally independent.
Time Frame: at 90 days post randomization
Population: The primary analysis was conducted according to intention to treat. All subjects were analyzed in the treatment group to which they were randomized. Subjects with missing mRS (n=9 in group two; n=4 in group one) or mRS assessed <60 days or >120 days post-randomization (n=10 in group two; n=4 in group one) are assigned an unfavorable outcome(mRS >2)
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants
  mRS 0-2 | 177 | 86
  mRS 3-6 | 257 | 136
Statistical Analysis 1: Comparison: Endovascular Therapy vs IV Rt-PA Alone; Test of null hypothesis (equal proportions of subjects with mRS of 0-2 at 90 days post-randomization in IV Only and Endovascular treatment arms) versus alternative hypothesis (unequal proportions of subjects with mRS of 0-2 at 90 days post-randomization in IV Only and Endovascular treatment arms); Test type: Superiority or Other; p = .7031, Cochran-Mantel-Haenszel — The CMH statistic is tested at the two-sided alpha level of 0.05. For the interim analyses of the primary efficacy analysis, the alpha spending function method (Lan and DeMets, 1987) with O'Brien and Fleming (1979) stopping boundaries were adopted; Cochran-Mantel-Haenszel (CMH) test adjusting for the dichotomized baseline NIHSS score (<20 or ≥20); Risk Difference (RD) = 1.5, 95% CI 2-sided [-6.1 to 9.1] — Positive adjusted risk difference indicates greater risk in the Endovascular group, while negative adjusted risk difference indicates greater risk in the IV Only group

2. Primary Outcome: Death Due to Any Cause
Time Frame: within 90 days post randomization
Population: The intent-to-treat analysis includes all subjects who were randomized, and each subject analyzed according to the treatment group to which they were randomly assigned. Subjects who ended the study prior to 90 days post- randomization for a reason other than death (LTFU etc) (n=8 in group two; n=2 in group one) are assumed to be alive
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants | 83 | 48
Statistical Analysis 1: Comparison: Endovascular Therapy vs IV Rt-PA Alone; Test of null hypothesis (equal proportions of subjects with mortality within 90 days post-randomization in IV Only and Endovascular treatment arms) versus alternative hypothesis (unequal proportions of subjects with mortality within 90 days post-randomization in IV Only and Endovascular treatment arms); Test type: Superiority or Other; p = .5241, Cochran-Mantel-Haenszel — The CMH statistic is tested at the two-sided alpha level of 0.01; Cochran-Mantel-Haenszel (CMH) test adjusting for the dichotomized baseline NIHSS score (<20 or ≥20); Risk Difference (RD) = -2.0, 99% CI 2-sided [-10.3 to 6.2] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Symptomatic Intracranial Hemorrhage
Description: Symptomatic Intracranial Hemorrhage- Symptomatic ICH is defined as an intracranial hemorrhage temporally related to a decline in neurological status as well as new or worsening neurologic symptoms in the judgment of the clinical investigator and which may warrant medical intervention. These events are identified via Adverse Event CRF submitted by the site
Time Frame: within the first 30 hours post IV rt-PA
Population: The intent-to-treat analysis sample includes all subjects who are randomized, and each subject is analyzed according to the treatment group to which they were randomly assigned.
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants | 27 | 13
Statistical Analysis 1: Comparison: Endovascular Therapy vs IV Rt-PA Alone; Test of null hypothesis (equal proportions of subjects with sICH within 30 hours post IV tPA initiation in IV Only and Endovascular treatment arms) versus alternative hypothesis (unequal proportions of subjects with sICH within 30 hours post IV tPA initiation in IV Only and Endovascular treatment arms); Test type: Superiority or Other; p = .8275, Cochran-Mantel-Haenszel — The CMH statistic is tested at the two-sided alpha level of 0.01; Cochran-Mantel-Haenszel (CMH) test adjusting for the dichotomized baseline NIHSS score (<20 or ≥20); Risk Difference (RD) = .4, 99% CI 2-sided [-4.6 to 5.5] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Incidence of Parenchymal Type II (PH2) Hematomas
Description: a dense intracerebral hematoma involving more than 30% of the infarcted area with substantial space-occupying effect or any hemorrhagic area outside the infarcted area, determined via central read of the submitted CT scans.
Time Frame: within 30 hours post IV rt-PA
Population: Subjects were excluded if a post-baseline CT scan was not obtained within 30 hours of randomization (i.e., participants who died, had care withdrawn at the request of the family, or underwent imaging after the 30-hour window).
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 417 | 207
participants | 25 | 13

5. Secondary Outcome: Asymptomatic Intracranial Hemorrhage
Description: Asymptomatic intracranial hemorrhage is defined as an intracranial hemorrhage without evidence of decline in neurological status or new or worsening neurologic symptoms in the judgment of the clinical investigator. These events are identified via Adverse Event CRF submitted by the site.
Time Frame: within 30 hours post IV rt-PA
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants | 119 | 42

6. Secondary Outcome: National Institutes of Health Stroke Scale Score (NIHSS) >> Dichotomized 0-1 Versus 2 or Greater.
Description: The National Institutes of Health Stroke Scale (NIHSS), a serial measure of neurologic deficit, is a 42-point scale that >> quantifies neurologic deficits in 11 categories, with 0 indicating normal function without neurologic deficit and higher
  >> scores indicating greater severity of deficit.
Time Frame: at 24 hours post randomization
Population: The intent-to-treat analysis sample includes all subjects who are randomized, and each subject is analyzed according to the treatment group to which they were randomly assigned. Subjects with missing NIHSS and NIHSS measured <18 hours or >30 hours post-randomization are assigned an unfavorable outcome (NIHSS score>1).
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants
  NIHSS 0-1 | 44 | 22
  NIHSS 2+ | 390 | 200

7. Secondary Outcome: National Institutes of Health Stroke Scale Score (NIHSS) Dichotomized 0-1 Versus 2 or Greater.
Description: The National Institutes of Health Stroke Scale (NIHSS), a serial measure of neurologic deficit, is a 42-point scale that quantifies neurologic deficits in 11 categories, with 0 indicating normal function without neurologic deficit and higher scores indicating greater severity of deficit.
Time Frame: at 90 days post randomization
Population: The intent-to-treat analysis sample includes all subjects who are randomized, and each subject is analyzed according to the treatment group to which they were randomly assigned. Subjects with missing NIHSS and NIHSS measured <60 days or >120 days post-randomization are assigned an unfavorable outcome (NIHSS score>1).
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants
  NIHSSS 0-1 | 120 | 50
  NIHSSS 2+ | 314 | 172

8. Secondary Outcome: Barthel Index (BI) Dichotomized 0-90 Versus 95-100
Description: The Barthel Index (BI)is an ordinal scale used to measure a subject's performance in activities of daily living (ADL) in ten variables- feeding, transfer (bed to chair), grooming, toilet use, bathing, mobility on a level surface, stair use, dressing, bowels and bladder. It is an assessment of independence in ADL and is scored in increments of 5 points. The lowest possible score on the index is 0 which implies total dependence on others for ADL and the highest total score is 100 which indicate full independent in ADL. A higher score is associated with a greater likelihood of being able to live at home with a degree of independence.
Time Frame: at 90 days post randomization
Population: The intent-to-treat analysis sample includes all subjects who are randomized, and each subject is analyzed according to the treatment group to which they were randomly assigned. Subjects with missing BI and BI measured <60 days or >120 days post-randomization are assigned an unfavorable outcome (BI 0-90).
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants
  BI 95-100 | 183 | 86
  BI 0-90 | 251 | 136

9. Secondary Outcome: Trail Making Test Part A Time
Description: The Trail Making Test is a neuropsychological test of visual attention and task switching that is thought to be sensitive to the presence of cerebral dysfunction. It is a timed test consisting of two parts where the subject is asked to draw a "trail" made by connecting numbers in sequential order (part A) and then in part B the combination of numbers and letters. Scoring is calculated separately for Parts A and B but both scores are provided as the minutes and seconds it takes for the subject to complete each part. Normally, the entire test (A and B) can be completed in 5 to 10 minutes.
Time Frame: 90 days post randomization
Population: Participants were excluded if the Trail Making Test was not assessed or if they failed to complete Part A.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 244 | 127
seconds | 84.2 (64.3) | 82.0 (62.3)

10. Secondary Outcome: Trail Making Test Part B Time
Description: as for outcome 9
Time Frame: at 90 days post randomization
Population: Participants were excluded if the Trail Making Test was not assessed or if they failed to complete Part B.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 183 | 92
seconds | 143.8 (75.3) | 141.3 (78.4)

11. Secondary Outcome: Modified Rankin Scale (mRS) Score Dichotomized to 0-2 Versus Greater Than 2
Description: as for outcome 1
Time Frame: at 180 days
Population: The intent-to-treat analysis sample includes all subjects who are randomized, and each subject is analyzed according to the treatment group to which they were randomly assigned. Subjects with missing mRS and mRS measured <150 days or >210 days post-randomization are assigned an unfavorable outcome (mRS>2).
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants
  mRS 0-2 | 179 | 86
  mRS 3-6 | 255 | 136

12. Secondary Outcome: Modified Rankin Scale (mRS) Score Dichotomized to 0-2 Versus Greater Than 2
Description: as for outcome 1
Time Frame: 270 days
Population: The intent-to-treat analysis sample includes all subjects who are randomized, and each subject is analyzed according to the treatment group to which they were randomly assigned. Subjects with missing mRS and mRS measured <240 days or >300 days post-randomization are assigned an unfavorable outcome (mRS>2).
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants
  mRS 0-2 | 177 | 88
  mRS 3-6 | 257 | 134

13. Secondary Outcome: Modified Rankin Scale (mRS) Score Dichotomized to 0-2 Versus Greater Than 2
Description: as for outcome 1
Time Frame: 360 days post randomization
Population: The intent-to-treat analysis sample includes all subjects who are randomized, and each subject is analyzed according to the treatment group to which they were randomly assigned. Subjects with missing mRS and mRS measured <330 days or >390 days post-randomization are assigned an unfavorable outcome (mRS>2).
Measure: Number; unit: participants
Arm/Group | Endovascular Therapy | IV Rt-PA Alone
Number analyzed (Participants) | 434 | 222
participants
  mRS 0-2 | 191 | 95
  mRS 3-6 | 243 | 127

ADVERSE EVENTS:
Groups:
- Endovascular: Group two will receive a lower dose or a standard dose of IV rt-PA and then undergo an angiogram test (cerebral angiography) rightafter the medicine is given to check for blood clots. If a clot is not seenthen no more treatment will be given. If a clot is seen, theneurointerventionalist will then choose (based on the location andextent of the blood clot) a protocol approved endovascular treatmentgiven directly in the brain artery that will be most effective inreopening the blocked artery.
- IV Only: Group one will receive the standard dose of intravenous (IV) rt-PA alone given over an hour.
Arm/Group | Endovascular | IV Only
Serious Adverse Events (participants affected / at risk) | 256/434 | 126/222
Other Adverse Events (participants affected / at risk) | 385/434 | 202/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=434) | IV Only (N=222)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 7 (8) | 5 (5)
Atrial flutter (Cardiac disorders) | 3 (3) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 8 (9) | 4 (4)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 4 (4)
Cardiac valve vegetation (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Electromechanical dissociation (Cardiac disorders) | 1 (1) | 0 (0)
Endocarditis noninfective (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 2 (2) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 4 (4)
Atrial septal defect (Congenital, familial and genetic disorders) | 4 (4) | 1 (1)
Hereditary cerebral degeneration (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Brain death (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 3 (4) | 0 (0)
Chest pain (General disorders) | 3 (3) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema due to cardiac disease (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 16 (17) | 8 (8)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 5 (5)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 8 (11) | 7 (7)
Urosepsis (Infections and infestations) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 7 (7) | 2 (3)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Difficult to wean from ventilator (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stent occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ventriculoperitoneal shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood osmolarity decreased (Investigations) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Computerised tomogram abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 1 (1)
Electroencephalogram abnormal (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
NIH stroke scale score increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Acid-base balance disorder mixed (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gliomatosis cerebri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Brain compression (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 46 (46) | 19 (20)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 3 (3) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 2 (2)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 8 (8) | 8 (8)
Cerebral infarction (Nervous system disorders) | 9 (9) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 18 (19) | 12 (12)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 9 (9) | 9 (9)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Facial spasm (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 12 (12) | 8 (8)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 6 (6) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 6 (7) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Neurological symptom (Nervous system disorders) | 12 (13) | 4 (4)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (2) | 0 (0)
Stroke in evolution (Nervous system disorders) | 0 (0) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 6 (6) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Emotional disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 6 (7) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 5 (5)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 2 (2) | 2 (3)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Craniectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cranioplasty (Surgical and medical procedures) | 9 (9) | 3 (3)
Intubation (Surgical and medical procedures) | 0 (0) | 1 (2)
Medical device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Tracheostomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial restenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 7 (7) | 2 (2)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 6 (6)
Iliac artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=434) | IV Only (N=222)
Anaemia (Blood and lymphatic system disorders) | 39 (41) | 16 (17)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 7 (7) | 5 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 4 (4) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 37 (41) | 21 (22)
Atrial flutter (Cardiac disorders) | 3 (4) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 18 (19) | 9 (9)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 16 (17) | 7 (8)
Cardiac valve disease (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac valve vegetation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 2 (2) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 7 (7)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 15 (16) | 9 (9)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 6 (6) | 3 (3)
Atrial septal defect (Congenital, familial and genetic disorders) | 3 (3) | 2 (2)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Homocystinaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (2) | 2 (2)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 2 (3) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Pupil fixed (Eye disorders) | 0 (0) | 1 (1)
Scleral oedema (Eye disorders) | 2 (2) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 41 (43) | 26 (27)
Diarrhoea (Gastrointestinal disorders) | 21 (21) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 14 (14) | 3 (3)
Faecal incontinence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 3 (3) | 6 (6)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 5 (5) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 43 (45) | 17 (18)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periproctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 39 (40) | 21 (22)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 3 (3) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 17 (17) | 9 (10)
Chills (General disorders) | 1 (1) | 1 (1)
Discomfort (General disorders) | 4 (4) | 1 (1)
Extravasation (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 2 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 10 (10) | 2 (2)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 4 (4) | 3 (3)
Hyperthermia (General disorders) | 0 (0) | 2 (2)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 1 (2) | 0 (0)
Infusion site haemorrhage (General disorders) | 4 (4) | 3 (3)
Infusion site oedema (General disorders) | 1 (1) | 0 (0)
Injection site extravasation (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 23 (29) | 13 (15)
Pain (General disorders) | 30 (32) | 14 (16)
Pitting oedema (General disorders) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 35 (36) | 31 (32)
Swelling (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1) | 1 (1)
Vessel puncture site haematoma (General disorders) | 15 (15) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 4 (4) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 2 (2) | 2 (2)
Fungal infection (Infections and infestations) | 5 (5) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion site infection (Infections and infestations) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 16 (16) | 6 (6)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 36 (39) | 8 (8)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 7 (7) | 2 (2)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subacute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 90 (104) | 46 (51)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 26 (30) | 9 (12)
Device lead damage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Difficult to wean from ventilator (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 13 (15) | 18 (18)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 5 (5) | 2 (3)
Incision site oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pacemaker complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 8 (9) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 4 (4) | 0 (0)
Bacteria stool identified (Investigations) | 1 (1) | 1 (1)
Blood albumin abnormal (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Blood culture positive (Investigations) | 0 (0) | 1 (1)
Blood electrolytes abnormal (Investigations) | 1 (1) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 8 (8) | 3 (3)
Blood phosphorus decreased (Investigations) | 2 (2) | 2 (2)
Blood potassium decreased (Investigations) | 2 (2) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 2 (2)
Blood test abnormal (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood urea abnormal (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 6 (6) | 2 (3)
Breath sounds abnormal (Investigations) | 1 (1) | 1 (3)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Chest X-ray abnormal (Investigations) | 0 (0) | 1 (1)
Computerised tomogram abnormal (Investigations) | 3 (3) | 1 (1)
Culture urine positive (Investigations) | 0 (0) | 1 (1)
Drug level fluctuating (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Electroencephalogram abnormal (Investigations) | 0 (0) | 1 (1)
Free prostate-specific antigen increased (Investigations) | 1 (1) | 0 (0)
Full blood count abnormal (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 3 (3) | 1 (1)
Haematology test abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin (Investigations) | 1 (1) | 0 (0)
Haemoglobin abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 8 (9) | 2 (2)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Inspiratory capacity decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Myoglobin blood increased (Investigations) | 1 (1) | 0 (0)
NIH stroke scale score increased (Investigations) | 1 (1) | 2 (2)
Neurological examination abnormal (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 3 (3) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0)
Residual urine volume (Investigations) | 1 (1) | 0 (0)
Scan with contrast abnormal (Investigations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 10 (10) | 3 (3)
Urine output decreased (Investigations) | 1 (1) | 2 (2)
Urine output increased (Investigations) | 1 (1) | 0 (0)
Venous pressure jugular increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 13 (13) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 23 (25) | 7 (7)
Fluid imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 31 (31) | 11 (11)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 10 (10)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (8) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 40 (40) | 18 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (14) | 7 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (25) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (24) | 13 (13)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 (18) | 8 (8)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (31) | 12 (17)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 3 (3) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 10 (10) | 15 (16)
Carotid arterial embolus (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 7 (8) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 5 (5) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 26 (26) | 7 (7)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 1 (2)
Cerebrovascular spasm (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 2 (2) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 16 (19) | 5 (5)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 3 (3) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 15 (17) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalomalacia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 43 (43) | 14 (14)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 35 (35) | 18 (18)
Headache (Nervous system disorders) | 80 (86) | 51 (55)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 2 (2)
Intention tremor (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 5 (6) | 5 (5)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 2 (2) | 1 (1)
Muscle spasticity (Nervous system disorders) | 3 (3) | 2 (2)
Neurological symptom (Nervous system disorders) | 12 (12) | 5 (5)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 5 (5) | 0 (0)
Partial seizures (Nervous system disorders) | 3 (3) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Putamen haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4) | 4 (4)
Subarachnoid haemorrhage (Nervous system disorders) | 8 (8) | 2 (2)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 1 (1)
Tremor (Nervous system disorders) | 5 (5) | 2 (2)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 31 (32) | 18 (19)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 24 (25) | 10 (11)
Bruxism (Psychiatric disorders) | 0 (0) | 1 (1)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 6 (6) | 0 (0)
Delirium (Psychiatric disorders) | 5 (5) | 1 (1)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 43 (44) | 18 (19)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 7 (7) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1)
Impulsive behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 26 (28) | 11 (11)
Insomnia related to another mental condition (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 4 (4) | 6 (7)
Osmophobia (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 3 (3) | 1 (1)
Posturing (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 3 (3) | 6 (6)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 24 (25) | 13 (13)
Hypertonic bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 2 (2) | 1 (1)
Oliguria (Renal and urinary disorders) | 6 (6) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 7 (7) | 2 (2)
Urinary retention (Renal and urinary disorders) | 13 (13) | 6 (7)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 10 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (2)
Tracheal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper airway resistance syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 5 (7) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (9)
Erythema (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Melanosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 17 (17) | 8 (8)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (4)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Drug abuser (Social circumstances) | 0 (0) | 1 (1)
Inadequate diet (Social circumstances) | 0 (0) | 1 (1)
Atrial septal defect repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cerebral oedema management (Surgical and medical procedures) | 2 (2) | 0 (0)
Cranioplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastrointestinal tube removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
High frequency ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral nerve decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Artery dissection (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 11 (11) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 14 (16) | 5 (6)
Haemorrhage (Vascular disorders) | 5 (5) | 0 (0)
Haemorrhagic infarction (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 30 (32) | 16 (16)
Hypotension (Vascular disorders) | 34 (34) | 23 (23)
Labile blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 3 (3) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 3 (3) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Vascular rupture (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The IMS III trial was stopped early because of futility, according to the prespecified rules. A limitation of our trial is that it did not compare the efficacy of the new stent retrievers with that of intravenous t-PA alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication will be authored prior to 12 mos after publication of the primary results without consent of the Publications Subcommittee. 12 mos after this time an Investigator may publish the results at the Collaborating Institution. No institution involved may be restricted from publishing independently 12 mos from publication of the primary paper. After 12 mo all manuscripts from the study must be submitted to the PI/Publications Subcommittee 45 days prior to any submission.